CLINICAL TRIAL: NCT04116801
Title: Evaluation of Resection Quality of Cerebral Metastases Using Fluorescence Guided Surgery: a Prospective Randomised Study- Fluomet Study
Brief Title: Evaluation of Resection Quality of Cerebral Metastases Using Fluorescence Guided Surgery: a Prospective Randomised Study
Acronym: Fluomet
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: Dr Philippe METELLUS (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-000515-16
Record Dates: First submitted 2019-10-03; First posted 2019-10-07 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Cerebral Metastases; Fluorescence Guided Surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluorescence arm (Experimental): fluorescence guided microsurgical resection (under 560 nm filter) in addition to the usual techniques, after iv injection of 200 mg (i.e. 3-4 mg/kg) of fluorescein sodium at the time of skin incision.
  Interventions: Procedure: microsurgical resection
- Standard excision (Active Comparator): microsurgical resection with usual techniques
  Interventions: Procedure: microsurgical resection

INTERVENTIONS:
Procedure: microsurgical resection — resection of cerebral metastases by microsurgery

SUMMARY:
Few studies have evaluated the use of fluorescein sodium for the resection of brain tumours (especially glioblastomas) but also cerebral metastases. We therefore propose to evaluate the technique of fluorescence guided microsurgery (fluorescein sodium) compared to the conventional microsurgical technique in the resection of cerebral metastases in adults in order to specify, by a prospective and randomised study, the assistance provided by this technique in the quality of resection and the gain in terms of overall survival and local control of brain disease.

DETAILED DESCRIPTION:
Cerebral metastases are a major public health problem in cancer patients. They are the most common brain tumours in adults. It is estimated that approximately 20-40% of patients with primary malignant neoplasia will develop cerebral metastasis during the course of their illness. In addition, the incidence of brain metastases is increasing due, in particular, to the aging of the population, as well as to the improvement of the overall management of cancer patients (cytotoxic or targeted systemic treatment) and easier access to magnetic resonance imaging (MRI), which improves patient survival. The prognosis of patients with brain metastases is still poor and the median overall survival of these patients is of the order of a few months. Although the management of brain metastases is multidisciplinary, the benefit of surgery has been clearly demonstrated in the literature. Consequently, it is demonstrated that the quality of the tumour excision and in particular the carrying out of the complete excision of contrast enhancement on the MRI is correlated with improved overall survival (especially in case of single metastasis) and improved local control of the disease or progression-free survival, but also a better quality of life. It is therefore essential to perform the most complete excision possible while minimising the associated morbidity. For this purpose, various tools for surgical resection have been developed and are available, including intraoperative fluorescence guided surgery. Sodium fluorescein is a fluorochrome that accumulates, after intravenous injection, into vascularised tumour tissues and is revealed intraoperatively by a light source of suitable wavelength (560 nm) using a set of lenses included in the microscope. The resection is thus guided by this fluorescence, the complete disappearance of which will translate into a complete tumour resection. Its interest is twofold: to increase the percentage of complete tumour resection and to improve survival without recurrence and overall survival.Few studies have evaluated the use of fluorescein sodium for the resection of brain tumours (especially glioblastomas) but also cerebral metastases. If two studies on brain metastases showed a complete resection rate greater than 80% and a better rate of local control of brain disease, it is important to note that these studies were not randomised (with a control arm), they did not really prove the effectiveness of this technique under fluorescence, hence the need to set up a randomised study. We therefore propose to evaluate the technique of fluorescence guided microsurgery (fluorescein sodium) compared to the conventional microsurgical technique in the resection of cerebral metastases in adults in order to specify, by a prospective and randomised study, the assistance provided by this technique in the quality of resection and the gain in terms of overall survival and local control of brain disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject over the age of 18 and under the age of 85
* Subject presenting 1 to 5 cerebral secondary locations of which one lesion (contrast enhancement of at least 1 cm) is accessible to the most complete excision possible
* Unprotected adult within the meaning of the law
* Subject belonging to a health insurance scheme
* Absence of medical contraindications to surgery and anaesthesia
* Absence of medical contraindications to performing an MRI
* Known absence of allergy to the injectable form of Fluorescein sodium
* Subject having signed their written informed consent.

Exclusion Criteria:

* Subject who is a minor, pregnant, parturient or breastfeeding woman
* Adult subject under legal protection, guardianship or deprivation of liberty by judicial or administrative decision
* Subject hospitalised without consent
* Anatomical localisation (cerebral trunk, diencephalon) of the cerebral metastasis counter-indicating a wide excision at the discretion of the neurosurgeon
* Subject participating in a clinical trial or any other research involving human beings
* Subject taking beta-blockers
* Subject who has not signed a written informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2017-09-19 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Quality excision | 48 hours
  To evaluate the quality of excision in both neurosurgical techniques, in terms of complete resection of cerebral metastases, objectified by the absence of quantifiable tumour residues on early postoperative MRI (before 48 hours) in both groups, evaluated by one of the neuroradiologists associated with the project.

CONTACTS AND LOCATIONS:
Locations (1):
- Clairval Private Hospital, Marseille, PACA, France

IPD SHARING:
Plan to Share IPD: Undecided